CLINICAL TRIAL: NCT05862857
Title: Innovative Strategies to Promote Biomedical HIV Prevention Uptake and Retention Among High-risk Adults at Drinking Venues in Kenya and Uganda
Brief Title: The Outreach and Prevention at ALcohol Venues in East Africa Study (OPAL-East Africa- Aim 1)
Acronym: OPAL-Aim 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Berkeley (Other); Makerere University (Other); Infectious Diseases Research Collaboration, Uganda (Other); Kenya Medical Research Institute (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-37054; 1R01AA030464-01 (NIH)
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: HIV/AIDS
Keywords: Drinking venues; Biomedical HIV prevention; Uganda; Kenya
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aim 1: HIV-focused mobilization (Active Comparator): Patrons and workers at drinking venues will be given a recruitment card for free HIV testing at the local clinic.
  Interventions: Behavioral: HIV-focused mobilization
- Aim 1: Multi-disease-focused mobilization (Experimental): Patrons and workers at drinking venues will be given a recruitment card for free multi-disease testing at the local clinic, including: diabetes, hypertension, HIV, malaria, TB, pregnancy.
  Interventions: Behavioral: Multi-disease-focused mobilization

INTERVENTIONS:
Behavioral: HIV-focused mobilization — Patrons and employees of drinking venues that are randomized to HIV-focused recruitment will receive a recruitment card offering free HIV testing at the local clinic
  Arms: Aim 1: HIV-focused mobilization
Behavioral: Multi-disease-focused mobilization — Patrons and employees of drinking venues that are randomized to HIV-focused recruitment will receive a recruitment card offering free health screenings that may include hypertension, diabetes, HIV, malaria (if febrile), and TB (if symptomatic), and pregnancy at the local clinic
  Arms: Aim 1: Multi-disease-focused mobilization

SUMMARY:
This study will test innovative interventions to increase uptake and use of biomedical HIV prevention options by engaging women and men at drinking venues in rural Kenya and Uganda in care, while gaining insights into the facilitators, barriers, and cost-effectiveness of these approaches.

DETAILED DESCRIPTION:
[BACKGROUND] Alcohol use is a common risk factor for both HIV prevention uptake and retention in sub-Saharan Africa (SSA). Interventions that promote biomedical HIV prevention (PrEP and PEP) among persons with heavy alcohol use and their sexual partners are urgently needed. Alcohol-serving drinking venues play an important role as sites of HIV transmission in SSA and are ideal sites to engage women and men at increased risk of HIV in biomedical prevention services.

[OVERVIEW] The investigators have developed a mobilization strategy of integrating HIV testing within multi-disease screening to recruit >2,000 people from drinking venues in Kenya and Uganda. The investigators now need to determine whether multi-disease mobilization can promote uptake of HIV prevention for adults at drinking venues in the context of new biomedical prevention options.

The project will rigorously test innovative interventions in Kenya and Uganda to increase uptake of biomedical HIV prevention, and assess facilitators, barriers, and cost-effectiveness of these approaches.

Specific Aims:

* Compare the effectiveness of two mobilization strategies to increase uptake of biomedical HIV prevention among adults at drinking venues.
* Determine the cost-effectiveness of interventions that increase biomedical HIV prevention uptake among adults at high-risk for HIV who attend drinking venues.

The proposed research will address the critical intersection of alcohol use and HIV risk in SSA, by promoting reach and uptake of biomedical HIV prevention and exploring associated facilitators and barriers.

ELIGIBILITY:
Participant Inclusion Criteria:

* adult (≥18 years)
* patron or worker at a drinking venue within the study community

Exclusion Criteria:

* age <18 years
* previous participation in the study (may only participate once)
* inability to consent (including gross inebriation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7727 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Biomedical HIV prevention uptake at 4 weeks | Measured 4 weeks after clinic screening visit
  The proportion of HIV-negative adults, receiving an Aim 1 recruitment card, who initiate PrEP or PEP after mobilization. This outcome will be measured by pill dispensing records and Ministry of Health (MoH) PrEP and PEP registry records.

SECONDARY OUTCOMES:
Biomedical HIV prevention uptake at 8 weeks | Measured 8 weeks after clinic screening visit
  The proportion of HIV-negative adults, receiving an Aim 1 recruitment card, who initiate PrEP or PEP after mobilization. This outcome will be measured by pill dispensing records and Ministry of Health (MoH) PrEP and PEP registry records.
Biomedical HIV prevention uptake at 12 weeks | Measured 12 weeks after clinic screening visit
  The proportion of HIV-negative adults, receiving an Aim 1 recruitment card, who initiate PrEP or PEP after mobilization. This outcome will be measured by pill dispensing records and Ministry of Health (MoH) PrEP and PEP registry records.
HIV testing uptake | Measured at clinic screening visit
  The proportion of HIV-negative adults, receiving an Aim 1 recruitment card, who accept clinic-based HIV testing at the clinic screening visit. HIV testing will be done in accordance with Kenyan and Ugandan national testing algorithms. Uptake will be recorded on study CRFs.
Yield of adults with untreated HIV | Measured at clinic screening visit
  The proportion of persons accepting HIV testing who are identified with newly diagnosed HIV or those who are self-reported to have known HIV infection but out of care and off of ART. HIV testing will be done in accordance with Kenyan and Ugandan national testing algorithms. Uptake, test results, HIV status, and current ART use will be recorded on study CRFs.
Yield of adults with heavy alcohol use | Measured at clinic screening visit
  Heavy alcohol use is defined as self-reported AUDIT-C score (a standardized, three question survey) of greater than or equal to 4 for men and greater than or equal to 3 for women. These outcomes will be recorded on study CRFs.
Adults with untreated HIV who initiate ART | Measured within one week of presenting for clinic-based screening with a recruitment card
  The proportion of adults with untreated HIV that initiate ART. Current and prior ART use will be self-reported and recoded on study CRFs. New ART prescriptions will be measured through pill dispensing data and MoH registries.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Chamie, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (2):
- Kenya Medical Research Institute (KEMRI), Mbita, Kenya
- Infectious Diseases Research Collaboration (IDRC), Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Per our Data Sharing agreement with the NIAAA Data Archive, we will share de-identified IPD from our baseline questionnaire, which includes questions about subject demographics, HIV risk, and alcohol use.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 3 months after article publication and the data will be made accessible for up to 36 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP).